CLINICAL TRIAL: NCT06779461
Title: A Prospective, Multicenter, Randomized, Open-Label, Parallel-Controlled Clinical Trial Assessing the Safety and Efficacy of Biodegradable Magnesium Embolic Microspheres for Primary Hepatocellular Carcinoma
Brief Title: A Clinical Trial Assessing the Safety and Efficacy of Biodegradable Magnesium Embolic Microspheres for Primary Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InnoBM Pharmaceuticals Co., Ltd. (Industry)
Collaborators: CHONGQING BAIMAITENGSHI PHARMACEUTICAL TECHNOLOGY CO., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BM601-Q001
Record Dates: First submitted 2024-12-25; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma Non-Resectable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cTACE (Placebo Comparator)
  Interventions: Procedure: cTACE
- cTACE with magnesium microspheres (Experimental)
  Interventions: Device: Magnesium Microspheres; Procedure: cTACE

INTERVENTIONS:
Device: Magnesium Microspheres — Biodegradable Magnesium Embolic Microspheres
  Arms: cTACE with magnesium microspheres
Procedure: cTACE — cTACE

SUMMARY:
The goal of this clinical trial is to determine if the addition of biodegradable magnesium metal microspheres to traditional TACE (Transarterial Chemoembolization) is effective in treating hepatocellular carcinoma, and to assess the safety of these microspheres.

The main questions it aims to answer are:

* Is the treatment more effective than traditional TACE alone?
* What additional medical issues arise when using the microspheres?

Researchers will compare TACE with magnesium microspheres to traditional TACE without microspheres to see if the addition of the microspheres improves treatment outcomes.

Participants will:

* Receive up to 3 treatments of TACE with or without microspheres
* Undergo checkups and tests every 30 days
* Keep records of tumor size and other safety issues

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 to 80 years inclusive, regardless of gender;
2. Patients with primary hepatocellular carcinoma (HCC) at CNLC stage Ib to IIIa who require transarterial chemoembolization (TACE) treatment and are unsuitable for or refuse surgical resection, liver transplantation, and ablation therapy;
3. ECOG score ≤ 2, and Child-Pugh classification of A or B;
4. Presence of at least one untreated, measurable tumor lesion with a diameter ≥ 3.0 cm according to mRECIST criteria (the maximum diameter of the target lesion ≤ 10.0 cm);
5. Patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) infection who are willing to receive antiviral treatment throughout the study period;
6. Voluntary participation in this clinical trial and signing of the informed consent form by the subject.

Exclusion Criteria:

1. Patients with prior embolization or other local treatments within 28 days before enrollment, or needing combined local treatment with TACE;
2. Received other antitumor systemic treatment within 28 days before enrollment;
3. Unsuitable for TACE due to lesion characteristics or vascular issues;
4. Vp3/Vp4 portal vein tumor thrombus;
5. Tumor occupying ≥70% of liver volume;
6. Decompensated cirrhosis or recent ascites drainage/TIPS;
7. Severe allergies to contrast agents or embolization materials;
8. Received blood products or certain corrective treatments within 7 days before enrollment;
9. Abnormal blood counts (WBC, platelets, neutrophils, hemoglobin);
10. Abnormal liver function tests (bilirubin, enzymes, albumin);
11. Renal impairment (creatinine, creatinine clearance);
12. Prolonged PT;
13. Unsuitable feeding artery for TACE or embolization risks;
14. Expected survival <6 months;
15. Pregnant, lactating, or planning pregnancy;
16. Factors affecting study results or necessitating study termination (alcoholism, drug abuse, severe diseases);
17. Severe infections unsuitable for TACE;
18. Participation in other clinical trials within 28 days before enrollment;
19. Other reasons deemed unsuitable by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ORR | 30 days after the last TACE treatment.
  The objective response rate of the target lesion

SECONDARY OUTCOMES:
Success rate of embolization technique for the target lesion | on the day of the surgery
  Success rate of embolization technique for the target lesion
DCR | 30 days after the first TACE treatment
  Disease control rate of the target lesion
CR | 30 days after the first TACE treatment
  Complete Response of the target lesion
ORR | 90 days after the last TACE treatment
  Objective Response Rate of the target lesion

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anyang Tumor Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Lishui Central Hospital, Lishui, Zhejiang
  - The Third Affiliated Hospital,Sun Yat-Sen University, Guangzhou
  - The First Hospital of Lanzhou University, Lanzhou
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No